CLINICAL TRIAL: NCT03694678
Title: Recovering Together: Building Resiliency in Dyads of Patients Admitted to the Neuroscience Intensive Care Unit (NICU) and Their Caregivers
Brief Title: Building Resiliency in Patients Admitted to the Neuroscience Intensive Care Unit and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Director of Integrated Brain Health Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018P002187
Record Dates: First submitted 2018-09-28; First posted 2018-10-03 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Acute Brain Injuries
Keywords: Psychiatry; Dyads; Patients; Caregivers; Psychosocial
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovering Together (Experimental): Dyads who are randomly assigned to the Recovering Together program will receive any usual clinic care as determined by their clinicians. Additionally, dyads will be invited to participate in 6 30-minute skills sessions. All sessions will include both pt and cg. A clinical psychologist will deliver the majority of sessions while the PI will deliver at least 10% of the sessions. The main intervention goal is to provide dyads with resiliency and interpersonal communication skills necessary to optimize their recovery and reduce emotional distress and PTS.
  Interventions: Behavioral: Recovering Together
- Health Education (No Intervention): Patients randomly assigned to the control condition will receive an educational program that mimics the dose and duration of the Recovering Together Program but without teaching any of the resiliency or interpersonal communication skills that are hypothesized to be responsible for improvement in emotional distress. The control will entail 2 in-person dyadic visits in the NICU and 4 dyadic virtual visits after discharge.

INTERVENTIONS:
Behavioral: Recovering Together — The intervention will teach resiliency skills (mindfulness, coping, interpersonal communication, etc) within 2 in person sessions at hospitalization and 4 live video sessions after discharge. Both patient and caregiver will participate in all sessions
  Arms: Recovering Together

SUMMARY:
The investigators will compare a dyadic intervention (Recovering Together) with an attention placebo educational control in dyads of patients with acute neurological illnesses and their caregivers at risk for chronic emotional distress. The primary aim of this study is to determine the feasibility, credibility, and satisfaction with Recovering Together. The second aim is to show proof of concept for sustained improvement in emotional distress, post traumatic stress (PTS), resiliency and interpersonal communication outcomes in patients and caregivers.

DETAILED DESCRIPTION:
The investigators aim to improve the care of patients (pts) admitted to the Neuroscience Intensive Care Unit (NICU) and their family caregivers (cgs) by conducting a pilot feasibility randomized controlled trial (RCT; N=80 dyads; 60 completers) of the dyadic resiliency program ("Recovering Together") to prevent chronic emotional distress in both pts and their cgs. Eligible dyads include adult, English speaking pts with acute neurological injury (ANI) admitted to the NICU, cleared medically and cognitively for participation by the nursing team, and their primary cgs. Dyads who are randomly assigned to "Recovering Together" will receive 6 manualized sessions (2 in person at hospitalization and 4 through live video after discharge, to reduce burden and facilitate access to care) led by a clinical psychologist. Dyads who are randomly assigned to the attention placebo educational control condition will receive 6 manualized sessions (2 in person and 4 through live video with a clinical psychologist), modeled after the Recovering Together program that will control for the dose of the intervention and support from therapist. Dyads will complete assessment surveys before, after the intervention and 3 months later. Clinical data on demographics, diagnosis, ANI severity, and any medical complications will be extracted from electronic health records.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 18 years or older
* English fluency and literacy
* Access to high speed internet for video sessions
* Patient with an informal cg (family or friend who provides unpaid care) available and willing to participate
* Hospitalized with an acute brain injury within 1-2 days when first approached, OR the primary caregiver of a patient currently admitted with an acute brain injury
* Either patient or caregiver within the dyads screens in for depression, anxiety, and/or PTSD

Exclusion Criteria:

* Permanent or severe cognitive impairment severe enough to impede participation - This will be determined by nurses through an assessment conducted as part of usual care (MMSE).
* Dyads where the patient is anticipated to die or to never be able to participate due to medical sequelae.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brasil S, de Carvalho Nogueira R, Salinet ASM, Yoshikawa MH, Teixeira MJ, Paiva W, Malbouisson LMS, Bor-Seng-Shu E, Panerai RB. Critical Closing Pressure and Cerebrovascular Resistance Responses to Intracranial Pressure Variations in Neurocritical Patients. Neurocrit Care. 2023 Oct;39(2):399-410. doi: 10.1007/s12028-023-01691-8. Epub 2023 Mar 3. PMID 36869208
- [Derived] Bannon SM, Cornelius T, Gates MV, Lester E, Mace RA, Popok P, Macklin EA, Rosand J, Vranceanu AM. Emotional distress in neuro-ICU survivor-caregiver dyads: The recovering together randomized clinical trial. Health Psychol. 2022 Apr;41(4):268-277. doi: 10.1037/hea0001102. Epub 2021 Sep 9. PMID 34498896
- [Derived] Vranceanu AM, Bannon S, Mace R, Lester E, Meyers E, Gates M, Popok P, Lin A, Salgueiro D, Tehan T, Macklin E, Rosand J. Feasibility and Efficacy of a Resiliency Intervention for the Prevention of Chronic Emotional Distress Among Survivor-Caregiver Dyads Admitted to the Neuroscience Intensive Care Unit: A Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2020807. doi: 10.1001/jamanetworkopen.2020.20807. PMID 33052404

RESULTS

PARTICIPANT FLOW:
Groups:
- Recovering Together: Dyads who are randomly assigned, via RedCap randomization, to the Recovering Together program received any usual clinic care as determined by their clinicians. Additionally, dyads were invited to participate in 6 30-minute skills sessions. All sessions included both pt and cg. A clinical psychologist delivered the majority of sessions while the PI delivered at least 10% of the sessions. The main intervention goal was to provide dyads with resiliency and interpersonal communication skills necessary to optimize their recovery and reduce emotional distress and PTS.
  Recovering Together: The intervention taught resiliency skills (mindfulness, coping, interpersonal communication, etc) within 2 in person sessions at hospitalization and 4 live video sessions after discharge. Both patient and caregiver participated in all sessions
- Health Education: Dyads who were randomly assigned, via RedCap randomization, to the control condition received an educational program that mimics the dose and duration of the Recovering Together Program but without teaching any of the resiliency or interpersonal communication skills that were hypothesized to be responsible for improvement in emotional distress. These sessions included health education content on self-care, including sleep, diet, movement, and exercise. The control entailed 2 in-person dyadic visits in the NICU and 4 dyadic virtual visits after discharge. Both patient and caregiver participated in all sessions.
Period: Overall Study
Arm/Group | Recovering Together | Health Education
Started (These numbers represent individual participants, not dyads.) | 60 | 62
Patient | 30 | 31
Caregiver | 30 | 31
Completed (Completers were participants who completed post-test. These numbers represent individual participants, not dyads.) | 56 | 59
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Population: Total number of participants (patients and caregivers) who completed >=1 intervention or control session were analyzed and included in baseline population.
Groups:
- Recovering Together: Patients; Recovering Together: Caregivers: Participants who are randomly assigned to the Recovering Together program received any usual clinic care as determined by their clinicians. Additionally, participants were invited to participate in 6 30-minute skills sessions. All sessions included both pt and cg. A clinical psychologist delivered the majority of sessions while the PI delivered at least 10% of the sessions. The main intervention goal was to provide dyads with resiliency and interpersonal communication skills necessary to optimize their recovery and reduce emotional distress and PTS.
  Recovering Together: The intervention taught resiliency skills (mindfulness, coping, interpersonal communication, etc) within 2 in person sessions at hospitalization and 4 live video sessions after discharge. Both patient and caregiver participated in all sessions
- Health Education: Patients; Health Education: Caregivers: Participants randomly assigned to the control condition received an educational program that mimics the dose and duration of the Recovering Together Program but without teaching any of the resiliency or interpersonal communication skills that were hypothesized to be responsible for improvement in emotional distress. The control entailed 2 in-person dyadic visits in the NICU and 4 dyadic virtual visits after discharge. All sessions included both pt and cg.
- Total: Total of all reporting groups
Arm/Group | Recovering Together: Patients | Recovering Together: Caregivers | Health Education: Patients | Health Education: Caregivers | Total
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Total number of participants (patients and caregivers) who completed >=1 intervention or control session were analyzed and included in baseline population.
  Years | 49.3 (16.7) | 52.4 (14.3) | 50.1 (16.4) | 52.1 (14.9) | 50.9 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Total number of participants (patients and caregivers) who completed >=1 intervention or control session were analyzed and included in baseline population.
  Participants
    Female | 9 | 22 | 12 | 17 | 60
    Male | 20 | 7 | 17 | 12 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total number of participants (patients and caregivers) who completed >=1 intervention or control session were analyzed and included in baseline population.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 1 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 2 | 4 | 2 | 3 | 11
    White | 25 | 25 | 24 | 20 | 94
    More than one race | 1 | 0 | 1 | 1 | 3
    Unknown or Not Reported | 0 | 0 | 1 | 4 | 5
Employment status [Count of Participants; unit: Participants]
  Employed full-time | 18 | 14 | 12 | 18 | 62
  Retired | 5 | 6 | 8 | 4 | 23
  Employed part-time | 1 | 3 | 1 | 2 | 7
  Homemaker | 0 | 2 | 1 | 2 | 5
  Full-time or part-time student | 1 | 1 | 1 | 1 | 4
  Other | 4 | 3 | 6 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment (Ability to Recruit Dyads)
Description: Feasibility of recruitment will be determined by reporting number of dyads who meet study criteria who enrolled
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: Approached participants who are eligible for the study
Arm/Group | Eligible Participants
Number analyzed (Participants) | 166
Participants
  Participants who enrolled and randomized | 122
  Participants who declined | 40
  Participants who enrolled and did not randomize | 4

2. Primary Outcome: Feasibility of Intervention Delivery (Ability to Deliver Intervention to Dyads)
Description: We will report number of sessions completed by each dyad. We will report any technical difficulties with live video delivery
Time Frame: Feasibility of program delivery will be measured at 6 weeks
Population: Number of dyads who started RT who had at least 1 member complete post treatment assessment
Measure: Number; unit: dyads
Groups:
- Health Education: Dyads randomly assigned to the control condition will receive an educational program that mimics the dose and duration of the Recovering Together Program but without teaching any of the resiliency or interpersonal communication skills that are hypothesized to be responsible for improvement in emotional distress. The control will entail 2 in-person dyadic visits in the NICU and 4 dyadic virtual visits after discharge.
Arm/Group | Recovering Together | Health Education
Number analyzed (Participants) | 30 | 31
dyads
  Number of dyads who started RT who had at least 1 member complete post treatment assessment | 29 | 31
  Number of dyads who started RT who had neither member complete post treatment assessment | 1 | 0

3. Primary Outcome: Credibility and Expectancy Questionnaire
Description: This measure will assess participants' belief that the intervention (or control) will be helpful. The score range is 3-27. Higher scores mean higher perception of credibility or expectancy.
Time Frame: Baseline
Population: Score on Credibility and Expectancy Questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovering Together | Health Education
Number analyzed (Participants) | 58 | 58
score on a scale
  Credibility and Expectancy Questionnaire; credibility subscale | 22.0 (4.4) | 20.3 (4.8)
  Credibility and Expectancy Questionnaire; expectancy subscale | 19.0 (5.2) | 19.5 (5.6)

4. Primary Outcome: Client Satisfaction Questionnaire
Description: This measure will assess participants' satisfaction with participation in the study. The score range is 0-12. Higher scores indicate greater satisfaction.
Time Frame: post intervention (6 weeks after baseline)
Population: Score on Client Satisfaction Questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovering Together | Health Education
Number analyzed (Participants) | 58 | 58
score on a scale | 10.65 (1.18) | 9.87 (2.70)

5. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: Measures symptoms of emotional distress and estimates diagnoses. The scale has 14 items, 7 assess anxiety and 7 depression. Scores range from 0-21 on each subscale, wtih higher scores indicating more symptoms. Scores greater than 8 indicate clinically significant symptoms.
Time Frame: baseline to posttest to 3 months follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Recovering Together: Patients: Patients whose dyad are randomly assigned to the Recovering Together program will receive any usual clinic care as determined by their clinicians. Additionally, dyads will be invited to participate in 6 30-minute skills sessions. All sessions will include both pt and cg. A clinical psychologist will deliver the majority of sessions while the PI will deliver at least 10% of the sessions. The main intervention goal is to provide dyads with resiliency and interpersonal communication skills necessary to optimize their recovery and reduce emotional distress and PTS.
  Recovering Together: The intervention will teach resiliency skills (mindfulness, coping, interpersonal communication, etc) within 2 in person sessions at hospitalization and 4 live video sessions after discharge. Both patient and caregiver will participate in all sessions
- Recovering Together: Caregivers: Caregivers whose dyad are randomly assigned to the Recovering Together program will receive any usual clinic care as determined by their clinicians. Additionally, dyads will be invited to participate in 6 30-minute skills sessions. All sessions will include both pt and cg. A clinical psychologist will deliver the majority of sessions while the PI will deliver at least 10% of the sessions. The main intervention goal is to provide dyads with resiliency and interpersonal communication skills necessary to optimize their recovery and reduce emotional distress and PTS.
  Recovering Together: The intervention will teach resiliency skills (mindfulness, coping, interpersonal communication, etc) within 2 in person sessions at hospitalization and 4 live video sessions after discharge. Both patient and caregiver will participate in all sessions
- Health Education: Patients: Patients whose dyad are randomly assigned to the control condition will receive an educational program that mimics the dose and duration of the Recovering Together Program but without teaching any of the resiliency or interpersonal communication skills that are hypothesized to be responsible for improvement in emotional distress. The control will entail 2 in-person dyadic visits in the NICU and 4 dyadic virtual visits after discharge.
- Health Education: Caregivers: Caregivers whose dyad are randomly assigned to the control condition will receive an educational program that mimics the dose and duration of the Recovering Together Program but without teaching any of the resiliency or interpersonal communication skills that are hypothesized to be responsible for improvement in emotional distress. The control will entail 2 in-person dyadic visits in the NICU and 4 dyadic virtual visits after discharge.
Arm/Group | Recovering Together: Patients | Recovering Together: Caregivers | Health Education: Patients | Health Education: Caregivers
Number analyzed (Participants) | 29 | 29 | 29 | 29
score on a scale
  Baseline: depression | 8.7 (4.2) | 7.8 (2.7) | 7.1 (4.0) | 4.8 (3.8)
  Posttreatment: depression | 4.0 (4.1) | 3.28 (3.37) | 7.2 (3.7) | 6.1 (5.4)
  3-month follow-up: depression | 3.7 (3.3) | 2.42 (2.58) | 7.7 (5.0) | 7.27 (5.28)
  Baseline: anxiety | 11.1 (4.7) | 13.2 (3.9) | 6.3 (4.0) | 7.0 (4.7)
  Posttreatment: anxiety | 3.3 (4.1) | 6.0 (3.8) | 8.5 (5.2) | 8.1 (6.1)
  3-month follow-up: anxiety | 4.7 (4.8) | 5.3 (3.8) | 8.9 (6.0) | 9.62 (5.02)

6. Secondary Outcome: Post Traumatic Checklist
Description: The PTSD CheckList - Civilian Version measures symptoms of post traumatic stress and determines diagnoses. Scores range from 17-85. Higher scores indicate more severe stress.
Time Frame: baseline to posttest to 3 months follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovering Together: Patients | Recovering Together: Caregivers | Health Education: Patients | Health Education: Caregivers
Number analyzed (Participants) | 29 | 29 | 29 | 29
score on a scale
  Baseline | 41.6 (12.9) | 43.2 (10.7) | 29.3 (12.1) | 29.4 (12.0)
  Posttreatment | 26.4 (10.8) | 39.3 (9.8) | 34.6 (12.1) | 35.9 (16.6)
  3-month follow-up | 28.2 (10.1) | 27.3 (7.7) | 41.7 (16.0) | 37.7 (16.1)

7. Secondary Outcome: Measures of Coping Style Part A
Description: The MOCS-A measures various coping strategies such as relaxation or adaptive thinking. Scores range from 0 to 52, and higher scores indicate greater self-perceived proficiency with these skills.
Time Frame: baseline to posttest to 3 months follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovering Together: Patients | Recovering Together: Caregivers | Health Education: Patients | Health Education: Caregivers
Number analyzed (Participants) | 29 | 29 | 29 | 29
score on a scale
  Baseline | 2.2 (.8) | 2.3 (.6) | 2.6 (.9) | 2.5 (.9)
  Posttest | 2.7 (.8) | 2.6 (1.1) | 2.4 (.8) | 2.4 (1.2)
  3-month follow-up | 2.5 (.7) | 2.5 (.9) | 2.2 (1.0) | 2.3 (1.0)

8. Secondary Outcome: Cognitive and Affective Mindfulness Scale Revised
Description: Measures mindfulness skills used in daily life. The scale ranges from 12 to 48 with higher scores indicating higher mindfulness.
Time Frame: baseline to post test to 3 months follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovering Together: Patients | Recovering Together: Caregivers | Health Education: Patients | Health Education: Caregivers
Number analyzed (Participants) | 29 | 29 | 29 | 29
score on a scale
  Baseline | 34.2 (7.0) | 34.6 (5.8) | 35.1 (7.8) | 36.4 (7.6)
  Posttreatment | 36.7 (7.7) | 36.3 (6.5) | 35.0 (10.7) | 36.7 (8.5)
  3-month follow-up | 35.5 (7.9) | 36.3 (7.5) | 32.3 (9.0) | 33.3 (9.4)

9. Secondary Outcome: Dyadic Relationship Scale
Description: The Dyadic Relationship Scale (DRS) has 2 sub scales that assess dyadic strains and dyadic positive interaction. Scales on each sub scale range from 1 to 4, with higher scores indicating great severity of the relevant construct.
Time Frame: Baseline, post treatment, 3-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovering Together: Patients | Recovering Together: Caregivers | Health Education: Patients | Health Education: Caregivers
Number analyzed (Participants) | 29 | 29 | 29 | 29
score on a scale
  Dyadic strain: baseline | 2.0 (.8) | 2.0 (.7) | 2.0 (.78) | 1.8 (.7)
  Dyadic strain: posttreatment | 1.6 (.6) | 2.01 (.8) | 2.0 (.9) | 2.1 (.9)
  Dyadic strain: 3-month follow-up | 1.9 (.8) | 2.2 (.8) | 2.0 (.9) | 2.2 (.8)
  Positive interactions: baseline | 3.1 (.5) | 3.0 (.5) | 3.2 (.6) | 3.3 (.4)
  Positive interactions: posttreatment | 3.4 (.6) | 3.3 (.5) | 2.97 (.77) | 3.2 (.7)
  Positive interactions: 3-month follow-up | 3.2 (.6) | 3.2 (.6) | 2.82 (.67) | 3.0 (.7)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Recovering Together: Patients: Patients who are randomly assigned to the Recovering Together program will receive any usual clinic care as determined by their clinicians. Additionally, patients and their caregivers will be invited to participate in 6 30-minute skills sessions. All sessions will include both pt and cg. A clinical psychologist will deliver the majority of sessions while the PI will deliver at least 10% of the sessions. The main intervention goal is to provide dyads with resiliency and interpersonal communication skills necessary to optimize their recovery and reduce emotional distress and PTS.
  Recovering Together: The intervention will teach resiliency skills (mindfulness, coping, interpersonal communication, etc) within 2 in person sessions at hospitalization and 4 live video sessions after discharge. Both patient and caregiver will participate in all sessions
- Recovering Together: Caregivers: Caregivers who are randomly assigned to the Recovering Together program will receive any usual clinic care as determined by their clinicians. Additionally, caregivers and their patients will be invited to participate in 6 30-minute skills sessions. All sessions will include both pt and cg. A clinical psychologist will deliver the majority of sessions while the PI will deliver at least 10% of the sessions. The main intervention goal is to provide dyads with resiliency and interpersonal communication skills necessary to optimize their recovery and reduce emotional distress and PTS.
  Recovering Together: The intervention will teach resiliency skills (mindfulness, coping, interpersonal communication, etc) within 2 in person sessions at hospitalization and 4 live video sessions after discharge. Both patient and caregiver will participate in all sessions
- Health Education: Patients: Patients randomly assigned to the control condition will receive an educational program that mimics the dose and duration of the Recovering Together Program but without teaching any of the resiliency or interpersonal communication skills that are hypothesized to be responsible for improvement in emotional distress. The control will entail 2 in-person dyadic visits in the NICU and 4 dyadic virtual visits after discharge.
- Health Education: Caregivers: Caregivers randomly assigned to the control condition will receive an educational program that mimics the dose and duration of the Recovering Together Program but without teaching any of the resiliency or interpersonal communication skills that are hypothesized to be responsible for improvement in emotional distress. The control will entail 2 in-person dyadic visits in the NICU and 4 dyadic virtual visits after discharge.
Arm/Group | Recovering Together: Patients | Recovering Together: Caregivers | Health Education: Patients | Health Education: Caregivers
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03694678/Prot_SAP_000.pdf